CLINICAL TRIAL: NCT06530121
Title: The Effect of Toolbox Training on Radiation Protection Practices of Health Professionals Working in Radioactive Areas
Brief Title: The Effect of Toolbox Training on Radiation Protection Practices of Health Professionals in Radioactive Workplaces
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Hatay Mustafa Kemal Univercity (Unknown); Turan Şahmaran (Unknown)
Responsible Party: Principal Investigator, Bircan Kara, Ph.d Lecturer, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: hmkubircankara
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Health Physics, Healthcare Professionals, Toolbox Trainings

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with experimental and control groups
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Toolbox trainings (Experimental): Training given with a single page material, lasting between 10-15 minutes, aimed at on-the-job application.
  Interventions: Behavioral: Toolbox trainings
- control group (No Intervention): uninterrupted and monitored group

INTERVENTIONS:
Behavioral: Toolbox trainings — Training given with a single page material, lasting between 10-15 minutes, aimed at on-the-job application.
  Arms: Toolbox trainings

SUMMARY:
This study will be conducted in a randomized controlled, pre-test, post-test and experimental group design to determine the effects of on-the-job training on radiation workers (radiation safety, protective clothing, awareness). The universe of the study was radiation workers using dosimeters at Hatay Mustafa Kemal University Health Practice and Research Hospital. The experimental group determined by randomization consisted of a total of 80 workers working in ionizing radiation departments. Data were collected with the Information Form, radiation safety and awareness Application Information Form (Pre-Test-Post-Test), radiation protection checklists and On-the-Job Training Evaluation Form. Descriptive statistical methods will be used in the evaluation of the data, independent sample t-test, dependent sample t-test will be used in the comparison of scores and the results of variance analysis in repeated measures will be used in the comparison of three follow-up scores.

DETAILED DESCRIPTION:
This study will be conducted in a randomized controlled, pre-test, post-test and experimental group design to determine the effects of on-the-job training on radiation workers (radiation safety, protective clothing, awareness). The universe of the study was radiation workers using dosimeters at Hatay Mustafa Kemal University Health Practice and Research Hospital. The experimental group determined by randomization consisted of a total of 80 workers working in ionizing radiation departments. Data were collected with the Information Form, radiation safety and awareness Application Information Form (Pre-Test-Post-Test), radiation protection checklists and On-the-Job Training Evaluation Form. Descriptive statistical methods will be used in the evaluation of the data, independent sample t-test, dependent sample t-test will be used in the comparison of scores and the results of variance analysis in repeated measures will be used in the comparison of three follow-up scores.

The risk of cancer increases when exposed to medium and high doses of radiation (0.1 - 0.2 Gy), however, it is not clear whether the risk of cancer increases with acute low doses (0.1 Gy or lower) or low dose rates (1). Cancer risk is directly related to the absorbed dose. Therefore, it is important to create a model to define the effects of low radiation dose on carcinogenicity. In the report published in 2019, UNSCEAR (United Nations Scientific Committee on the Effects of Atomic Radiation) stated that the dose distributions and results arising from occupational exposure provide information about the source and conditions of exposure (2). This information has shown that the problems arising from radiation in departments working with ionizing radiation should be determined and further investigated. In addition, the protection of health professionals working in radioactive areas from radiation is important for both employee health and patient health. In particular, the implementation of the standards required for protection from radiation will emerge in this context and will provide protection from personal and institutional harm. In this context, it is very important for health professionals to address this issue more effectively in in-service training. In addition, it is thought that the time allocated by employees in environments such as hospitals, where the workload is high and the patient density is quite high, is quite limited and these personnel have little interest in in-service training provided with mass training methods. In this context, it is suggested that providing training to personnel with new training methods in environments such as hospitals will increase the permanence and impact of the training.

It is thought that this study will reveal the effects of new training methods on radiation protection practices of health workers working in radioactive areas, apart from mass training methods and routinely provided classical training methods, and will provide evidence for the use of this training method in addition to classical training methods.

10. Purpose of the study: The purpose of this randomized controlled, pre-test, post-test and experimental group design study is to provide on-the-job training to radiation officers working at Hatay Mustafa Kemal University Health Practice and Research Hospital and to investigate the effects of on-the-job training on radiation safety practices.

Place of the study: Hatay Mustafa Kemal University Health Practice and Research Hospital Universe and sample: The sample size of this study was determined using the simple random (randomized controlled) sampling method. It is planned to assign a total of 8 radioactive field workers who meet the sampling inclusion criteria to the experimental and control groups by drawing lots among the areas they work with the help of an external expert. It is planned that there will be a total of 80 radioactive field workers in the experimental and control groups to be assigned to the experimental and control groups as a result of the drawing lots, and 40 of this number will constitute the experimental group and 40 will constitute the control group.

Inclusion criteria:

* Working in radioactive areas
* Being a health professional
* Accepting to participate in the study voluntarily
* Working for at least 6 months

  12. The method planned to be used in the study: The universe of this study will consist of healthcare workers working in the radioactive areas of Hatay Mustafa Kemal University Health Practice and Research Hospital. The sample size of this study was determined using the simple random randomized controlled sampling method. It is planned to assign healthcare workers who meet the sampling inclusion criteria to experimental and control groups by drawing lots with the help of an external expert. According to the drawing results, experimental and control groups will be determined and on-the-job training will be given to the experimental group and radiation safety practices will be observed.

It is thought that this study will reveal the effects of new training methods other than mass training methods and routinely provided classical training methods on radiation protection practices of healthcare workers working in radioactive areas and will provide evidence for the use of this training method in addition to classical training methods.

Purpose of the study: The purpose of this randomized controlled, pre-test, post-test and experimental group design study is to provide on-the-job training to radiation officers working at Hatay Mustafa Kemal University Health Practice and Research Hospital and to investigate the effects of on-the-job training on radiation safety practices.

ELIGIBILITY:
Inclusion Criteria:

* Working in radioactive areas
* Being a health professional
* Agreeing to participate in the study voluntarily
* Working for at least 6 months

Exclusion Criteria:

* Working in any field other than radioactive areas
* Not being a health professional
* Working less than 6 months

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-08-28 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
pretest-posttest | before education and 1st week after training
  It consists of 10 multiple choice questions created to measure the knowledge levels of the participants before and after the training.

SECONDARY OUTCOMES:
radiation protection practices checklist | pre-training and post-training 1st week
  Applications that form the basis of radiation protection applications consisting of 8 items

IPD SHARING:
Plan to Share IPD: Yes
The research results will be reported and shared with researchers after the research is completed.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: will be published in the article together with the research results

REFERENCES:
- [Derived] Kara B, Sahmaran T. Evaluating the Impact of Toolbox Training on Health Professionals in Radiation Environments: A Randomized Controlled Trial. Health Phys. 2026 Mar 1;130(3):342-354. doi: 10.1097/HP.0000000000002101. Epub 2026 Jan 28. PMID 41631967